#### **SUMMARY OF CHANGES**

NCI Protocol #: 10212 Local Protocol #: OSU 18296

NCI Version Date: March 26, 2019 Protocol Date: March 26, 2019

### I. NCI Rapid Request Amendment (RRA) 03/26/2019

| # | Section | Page(s) | Change |
|---|---|---|---|
| 1. | <u>Header</u> | All | Updated Header Version Date to match updated protocol version |
| 2. | What risks, side effects or discomforts can my child expect from being in the study? | 2 | <ul> <li>Updated risks for pinometastat, per the revised condensed risk profile based on CAEPR (Version 1.1, January 7,2019)</li> <li>Added New Risk: <ul> <li>Possible: Diarrhea, nausea, vomiting; Tiredness; Change in the heart rhythm; Rash</li> </ul> </li> <li>Increase in Risk Attribution: <ul> <li>Changed to Possible from Also Reported on Pinometostat Trials But With Insufficient Evidence for Attribution (i.e., added to the Risk Profile): Anemia which may require blood transfusion; Bruising, bleeding</li> </ul> </li> <li>Decrease in Risk Attribution: <ul> <li>Changed to Also Reported on Pinometostat Trials But With Insufficient Evidence for Attribution from Possible (i.e., removed from the Risk Profile): Constipation; Severe blood infection; Bleeding in the brain which may cause headache, confusion</li> </ul> </li> </ul> |

## Parental Permission Authorization for Child's Participation in Research

**Study Title for Participants:** Testing the addition of a new anti-cancer drug, pinometostat, to the usual chemotherapy treatment (cytarabine and daunorubicin) in patients with Acute Myeloid Leukemia

Official Study Title for Internet Search on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>: "NCI-10212: A Phase 1b/2 study of Pinometostat in combination with standard induction chemotherapy in newly diagnosed Acute Myeloid Leukemia with MLL rearrangement," (NCT#PENDING)

- This is a parental permission form for research participation. It contains important information about this study and what to expect if you permit your child to participate. Please consider the information carefully. Feel free to discuss the study with your friends and family and to ask questions before making your decision whether or not to permit your child to participate.
- Your child's participation is voluntary. You or your child may refuse participation in this study. If your child takes part in the study, you or your child may decide to leave the study at any time. No matter what decision you make, there will be no penalty to your child and neither you nor your child will lose any of your usual benefits. Your decision will not affect your future relationship with The Ohio State University. If you or your child is a student or employee at Ohio State, your decision will not affect your grades or employment status.
- Your child may or may not benefit as a result of participating in this study. Also, as explained below, your child's participation may result in unintended or harmful effects for him or her that may be minor or may be serious depending on the nature of the research.
- You and your child will be provided with any new information that develops during the study that may affect your decision whether or not to continue to participate. If you permit your child to participate, you will be asked to sign this form and will receive a copy of the form. You are being asked to consider permitting your child to participate in this study for the reasons explained below.

### 1. Why is this study being done?

This study is being done to answer the following question:

Can we increase the chance of better treating AML by adding a new drug to the usual combination of drugs?

We are doing this study because we want to find out if this approach is better or worse than the usual approach for your AML. The usual approach is defined as care most people get for AML.

#### 2. How many people will take part in this study?

There will be about 6-37 people taking part in this study

#### 3. What will happen if my child takes part in this study?

If your child participates in this study, they will get Pinometostat for up to 35 days, in combination with standard intensive induction chemotherapy.

After your child finishes their 35 days of pinometostat, the doctor will continue to follow their condition and watch them for side effects. The follow up will occur either until their AML comes back or worsens, or until they get a different treatment for their AML. The follow up will occur during regular clinic visits with their hematologist at least every month.

Your child may choose to participate in an optional research bone marrow aspiration and biopsy to be performed on Day 8, where 1 teaspoon of blood and 1 teaspoon of bone marrow aspirate would be collected from them for research purposes only.

### 4. Can my child stop being in the study?

You child may stop being in the study at any time.

If they decide to stop, they should let the study doctor know as soon as possible. It's important that they stop safely. If they stop, they can decide if they want to keep letting the study doctor know how they are doing.

Their study doctor will tell them about new information or changes in the study that may affect their health or their willingness to continue in the study.

## 5. What risks, side effects or discomforts can my child expect from being in the study?

Your child may experience side effects from the pinometostat which include:

- Anemia which may require blood transfusion
- Infection, especially when white blood cell count is low
- Heart Failure, which may cause shortness of breath, swelling of ankles, and tiredness
- Diarrhea, nausea, vomiting
- Tiredness
- Change in the heart rhythm
- Bruising, Bleeding
- Rash

Your child may also experience side effects from their usual care:

- Diarrhea, loss of appetite, nausea, vomiting
- Anemia
- Fever
- Rash
- Blood clots

Mouth Sores

Your child may experience side effects from the bone marrow collection:

- Small amount of bleeding
- Bruising
- Pain

#### Risks to an unborn child or a baby:

If your child is a female it is important that they do not get pregnant or breastfeed a baby while participating in this study (at least 4 weeks after their last dose of study treatment). If your child is a male it is important that they do not father a baby while taking part in this study (at least 90 days after their last dose of study treatment).

### 6. What benefits can my child expect from being in the study?

This study drug has shrunk or stabilized your child's type of cancer in a limited number of people with their type of cancer. It is unlikely that it will work in everyone with their type of cancer or help you live longer. This study may help the study doctors learn things that may help other people in the future.

## 7. What other choices does my child have if he/she does not take part in the study?

- They may choose to have the usual approach described above.
- They may choose to take part in a different research study, if one is available.
- They may choose not to be treated for cancer.
- They may choose to only get comfort care to help relieve your symptoms and not get treated for your cancer.

### 8. What are the costs of taking part in this study?

You and/or your insurance plan will need to pay for the costs of medical care you get as part of the study, just as you would if you were getting the usual care for your AML. This includes:

- The costs of tests, exams, procedures, and drugs that you get during the study to monitor your safety, and prevent and treat side effects.
- The costs of daunorubicin and cytarabine.
- Your insurance co-pays and deductibles.

Talk to your insurance provider and make sure that you understand what your insurance pays for and what it doesn't pay for if you take part in this clinical trial. Also, find out if you need approval from your plan before you can take part in the study.

Ask your doctor or nurse for help finding the right person to talk to if you are unsure which costs will be billed to you or your insurance provider.

You and/or your insurance provider will not have to pay for exams, tests, and procedures done for research purposes only or that are covered by the study. These include:

- Bone marrow aspiration and biopsy done before treatment
- Bone marrow aspiration and biopsy done at relapse (if applicable)
- Bone marrow aspiration on day 8, and the genetic and chemical tests done on this specimen

You or your insurance provider will not have to pay for the Pinometostat while your child takes part in this study.

You and your child will not be paid for taking part in this study. The research may lead to new tests, drugs, or other products for sale. If it does, you will not get any payment.

#### 9. Will I or my child be paid for taking part in this study?

You and your child will not receive any payments or reimbursements for participating in this study.

# 10. What happens if my child is injured because he/she took part in this study?

If your child is injured as a result of taking part in this study and need medical treatment, please talk with their study doctor right away about their treatment options. The study sponsors will not pay for medical treatment for injury. Your insurance company may not be willing to pay for a study-related injury. Ask them if they will pay. If you do not have insurance, then you would need to pay for these medical costs.

If you feel this injury was caused by medical error on the part of the study doctors or others involved in the study, you have the legal right to seek payment, even though your child is in a study. Agreeing to take part in this study does not mean you or your child give up these rights.

### 11. What are my child's rights if he/she takes part in this study?

If you and your child choose to participate in the study, you and your child may discontinue participation at any time without penalty or loss of benefits. By signing this form, you do not give up any personal legal rights your child may have as a participant in this study.

You and your child will be provided with any new information that develops during the course of the research that may affect your decision whether or not to continue participation in the study.

You and your child may refuse to participate in this study without penalty or loss of benefits to which they are otherwise entitled.

### 12. Will my child's study-related information be kept private?

Your child's privacy is very important to us. The study doctors will make every effort to protect it. The study doctors have a privacy permit to help protect your child's records if there is a court case. However, some of their medical information may be given out if required by law. If this

should happen, the study doctors will do their best to make sure that any information that goes out to others will not identify who they are.

Some of your child's health information, such as their response to cancer treatment, results of study tests, and medicines they took, will be kept by the study sponsor in a central research database. However, their name and contact information will not be put in the database. If information from this study is published or presented at scientific meetings, their name and other personal information will not be used.

There are organizations that may look at your child's study records. Their health information in the research database also may be shared with these organizations. They must keep your child's information private, unless required by law to give it to another group. Some of these organizations are:

- The study sponsor and any drug company supporting the study
- The IRB, which is a group of people who review the research with the goal of protecting the people who take part in the study.
- The FDA and the groups it works with to review research
- The NCI and the groups it works with to review research.
- The NCI's National Clinical Trials Network and the groups it works with to conduct research

Your child's study records also will be stored for future use. However, their name and other personal information will not be used. Some types of future research may include looking at their records and those of other patients to see who had side effects across many studies or comparing new study data with older study data. However, we don't know what research may be done in the future using their information. This means that:

You and your child will not be asked if they agree to take part in the specific future research studies using their health information.

You and your child and their study doctor will not be told when or what type of research will be done. You and your child will not get reports or other information about any research that is done using your information.

There are laws that protect your child's genetic information. However, there is a risk that someone could get access to their genetic information and identify them by name. In some cases, employers could use their genetic information to decide whether to hire or fire them. The study doctors believe the risk of this happening is very small. However, the risk may increase in the future as people find new ways of tracing information. For more information about the laws that protect your child, ask your child's study doctor.

## **13. Who may use and give out information about your child?** Researchers and study staff.

### Signing the parental permission form

I have read (or someone has read to me) this form and I am aware that I am being asked to provide permission for my child to participate in a research study. I have had the opportunity to ask questions and have had them answered to my satisfaction. I voluntarily agree to permit my child to participate in this study.

I am not giving up any legal rights by signing this form. I will be given a copy of this combined consent and HIPAA research authorization form.

| Printed name of subject | |
|---|---|
| Printed name of person authorized to provide permission for subject | Signature of person authorized to provide permission for subject |
| | AM/PM |
| Relationship to the subject | Date and time |
| If your child is participating in the optional Day from an additional person authorized to provide | |
| Printed name of an additional person authorized to provide permission for subject | Signature of an additional person authorized to provide permission for subject |
| Relationship to the subject | Date and time |
| Investigator/Research Staff | |
| I have explained the research to the participant or h signature(s) above. There are no blanks in this doct the participant or his/her representative. | |
| Printed name of person obtaining consent | Signature of person obtaining consent |
| - | A 3.6 (D3.6 |
| | Date and time AM/PM |

### Witness(es) - May be left blank if not required by the IRB

| Printed name of witness | Signature of witness | |
|-------------------------|----------------------|-------|
| | | AM/PM |
| | Date and time | |
| Printed name of witness | Signature of witness | |
| Timed name of witness | Signature of witness | |
| | | AM/PM |
| | Date and time | |